CLINICAL TRIAL: NCT00730262
Title: A Phase II Study of TLN-4601 in Patients With Glioblastoma Multiforme
Brief Title: Efficacy Study of TLN-4601 in Patients With Recurring Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Thallion Pharmaceuticals (Industry)
Responsible Party: Didier Reymond, MD / Vice-President Medical and Clinical Affairs, Thallion Pharmaceuticals Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLN-4601-201
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme (GBM); Phase II; Brain Cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — diazepinomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm (Experimental)
  Interventions: Drug: TLN-4601

INTERVENTIONS:
Drug: TLN-4601 — 14 day continuous IV administration of TLN-4601 at 480 mg/m2/day followed by a 7-day recovery period
  Other Names: Formerly ECO-4601

SUMMARY:
The objective of this study is to assess the efficacy and safety of TLN-4601 used to treat patients with Glioblastoma Multiforme(GBM) that recur/progress after receiving first line systemic therapy post surgery/radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Glioblastoma Multiforme (GBM)
* Prior treatment with radiation and one first line systemic therapy (including temozolomide or other chemotherapy, immunotherapy, targeted therapy or combination therapies), followed by measurable and unequivocal evidence of tumor progression or recurrence
* Age ≥ 18 years
* ECOG ≤ 2
* Normal organ and marrow function as defined below:

  * leukocytes ≥3 x 109/L
  * absolute neutrophil count ≥1.5 x 109/L
  * platelets ≥100 x 109/L
  * hemoglobin ≥90 g/L
  * total bilirubin ≤2.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * creatinine ≤1.0 X institutional upper limit of normal

Exclusion Criteria:

* Patients with a life expectancy < 12 weeks
* Patients with a documented history of HIV, active hepatitis B or C infections
* Female patients who are pregnant or lactating
* Patients in whom a proper central line (Portacath-like device) cannot be established
* Patients with a known hypersensitivity to farnesylated dibenzodiazepinone or polysorbate 80
* Patients with uncontrolled hypotension
* Patients with concomitant therapy of therapeutic coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-04 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of TLN-4601 in patients with recurrent glioblastoma multiforme (GBM) as measured by 6-month progression free survival from date of initial infusion of TLN-4601 (Day 1, Cycle 1). | 6-month progression free survival from date of initial infusion of TLN-4601 (Day 1, Cycle 1)

SECONDARY OUTCOMES:
To examine the safety and tolerability of TLN-4601 in patients with recurrent GBM | Maximum 13 months from date of initial infusion of TLN-4601 (Day 1, Cycle 1)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Mason, MD, Principal Investigator — The Pencer Brain Tumor Center, Princess Margaret Hospital, Toronto
Locations (8):
- United States (2):
  - Sloan-Kettering Institute for Cancer Research, New York, New York
  - Duke University, Durham, North Carolina
- Canada (6):
  - Ottawa Health Research Institute, Ottawa, Ontario
  - The Pencer Brain Tumor Center, Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Notre-Dame du CHUM, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - L'Hotel-Dieu de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec